CLINICAL TRIAL: NCT06356181
Title: High-Intensity Functional Training Adaptations With and Without Maximus Ventilatory Training Device
Brief Title: Training Adaptations With and Without Ventilatory Training Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: MAXIMUS (Unknown)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor and Chair of Exercise Science Department, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00135143
Record Dates: First submitted 2024-03-27; First posted 2024-04-10 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: high-intensity functional training; respiratory training device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants in this group will undergo 6 weeks of high-intensity functional training using the respiratory muscle training device.
  Interventions: Device: Respiratory Maximus Training Device
- Control (Active Comparator): Participants in this group will undergo 6 weeks of high-intensity functional training without using the respiratory muscle training device.
  Interventions: Device: No Respiratory Training Device

INTERVENTIONS:
Device: Respiratory Maximus Training Device — Those in the intervention group will wear the respiratory training device for 3 days per week of high-intensity functional training over 6-weeks.
  Arms: Experimental
Device: No Respiratory Training Device — Those in the control group will train for 3 days per week of high-intensity functional training over 6-weeks.
  Arms: Control

SUMMARY:
This project aims to assess the effectiveness of using a Respiratory Muscle Training (RMT) device during high-intensity functional training (HIFT) to improve fitness and ventilatory parameters. Primary outcome measures include aerobic, anaerobic, and HIFT measures. Secondary measures include sleep, affect, and mood state questionnaires. Participants will be randomized into one of two groups: with the RMT device and without the RMT device.

DETAILED DESCRIPTION:
This study assesses the impact of a ventilatory training device, similar to a sports mouth guard worn during exercise, on various performance outcomes. The main questions it aims to answer are:

* Does the device improve fitness parameters: high-intensity functional training, anaerobic capacity, anaerobic peak and mean power output, maximal oxygen uptake, ventilatory threshold, and blood lactate responses to training?
* Does the device improve spirometry measures?

Researchers will compare 6 weeks of training with the ventilatory training device to those without the training device.

Participants will:

* Take part in a total of 8 weeks of study-related activity.
* Complete six total one- to two-hour pre- and post-testing sessions, which include a maximal oxygen uptake test, high-intensity functional training, body composition, spirometry, anaerobic power and capacity testing.
* Complete six weeks of 45-minute high-intensity functional training, three days per week.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 35 (inclusive) who participate in at least 150 minutes per week of physical activity.
* Have not participated in HIFT training in the last 6 months.
* Provided written and dated informed consent to participate in the study.
* In good health as determined by medical history and is cleared for exercise.
* Participant will be asked about dietary supplementation use within the past 6 months.

  * If participant began taking a supplement within the past month, subject will be asked to discontinue supplement use followed by a 2-week washout prior to participation.
  * In all other cases, we will request that participant maintain supplement use.

Exclusion Criteria:

* Any musculoskeletal injuries that would prevent exercising.
* Any metabolic disorder including known electrolyte abnormalities, diabetes, uncontrolled thyroid disease, adrenal disease or hypogonadism.
* Any inborn error of metabolism.
* History of hepatorenal, musculoskeletal, autoimmune, or neurologic disease.
* Participants with a personal history of heart disease, high blood pressure (systolic >140 mm Hg & diastolic >90 mm Hg),
* Participants who are pregnant, planning to become pregnant, or lactating.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Changes in spirometry | Baseline and Week 8
  Spirometry measures of forced vital capacity (FVC) (L), forced expiratory volume at one second (FEV1) (L), and the ratio of FEV1/FVC %
Changes in aerobic capacity | Baseline and Week 8
  Assessed via a cycle-ergometer based maximal graded exercise test with indirect calorimetry.
Changes in peak power | Baseline and Week 8
  Assessed via a cycle-ergometer based maximal graded exercise test
Changes in ventilatory threshold | Baseline and Week 8
  Assessed via a cycle-ergometer based maximal graded exercise test with indirect calorimetry.
Changes in countermovement jump | Baseline and Week 8
  Assessed via force plates
Changes in anaerobic capacity | Baseline and Week 8
  Assessed via 30-second Wingate test.
Changes in high-intensity functional training test | Baseline and Week 8
  Assessed via a high-intensity functional training circuit composed of rows, pushups, and squats
Changes in heart rate at ventilatory threshold | Baseline and Week 8
  Assessed via a cycle-ergometer based maximal graded exercise test with indirect calorimetry.

SECONDARY OUTCOMES:
Changes in body composition | Baseline and Week 8
  Body fat percentage, fat-free mass, and fat mass via air-displacement plethysmography.
Changes in sleep quality | Baseline and Weeks 3, 5, and 7
  Assessed by Pittsburgh Sleep Quality Index. The minimum score is 0 and the maximum score is 40. Higher scores mean a worse outcome.
Changes in total mood disturbances | Baseline and Weeks 3, 5, and 7
  Assessed by the Profile of Mood States (POMS). The total mood is calculated by adding the negative subscales (tension, depression, fatigue, confusion, and anger) and subtracting the positive subscales (vigor, esteem-related affect). Minimum score of -36 and max score of 200. Lower scores for total mood disturbance are considered better.
Changes in positive mood and emotion | Baseline and Weeks 3, 5, and 7
  Assessed by the Positive and Negative Affect Schedule. Min values of 0 and max of 50, higher scores indicate more positive moods and emotions.
Change in blood lactate responses | Weeks 3, 5, and 7
  Biochemical responses to exercise. Blood lactate sampled pre and post exercise during the last training day of the week.
Changes in negative mood and emotion | Baseline and Weeks 3, 5, and 7.
  Assessed by the Positive and Negative Affect Schedule. Min values of 0 and max of 50, higher scores indicate more negative moods and emotions with lower scores indicating less negative moods and emotions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No